CLINICAL TRIAL: NCT02051764
Title: An Open Label, Multicenter Study, Evaluating the Imaging Characteristics of a Follow-up 18F-AV-1451 Scan in Subjects Who Have Had a Prior 18F-AV-1451 Scan
Brief Title: Imaging Characteristics of a Follow-up 18F-AV-1451 Scan
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lower than expected enrollment
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A04
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Follow-up Flortaucipir PET Scan (Experimental)
  Interventions: Drug: Flortaucipir F18; Drug: Florbetapir F 18; Procedure: Brain PET Scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: 18F-AV-1451; LY3191748; [F-18]T807
Drug: Florbetapir F 18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: Amyvid; 18F-AV-45
Procedure: Brain PET Scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This study will evaluate the imaging characteristics of flortaucipir in subjects with a previous flortaucipir scan in order to assess the rate of change of tau deposition over time.

ELIGIBILITY:
Inclusion Criteria:

* Have a previous 18F-AV-1451 brain scan
* Can tolerate up to two Positron Emission Tomography (PET) imaging sessions and a Magnetic Resonance Imaging (MRI) scan
* Ability to provide informed consent

Exclusion Criteria:

* Current clinically significant psychiatric disease
* Are claustrophobic
* Current clinically significant cardiovascular disease or ECG abnormalities, or additional risk factors for Torsades de Pointes
* Current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Hoag Memorial Hospital, Newport Beach, California
  - UC Irvine Medical Center, Orange, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Center for Clinical Imaging Research, Washington University School of Medicine, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled subjects who had previously undergone flortaucipir PET (positron emission tomography) scans in other Avid-sponsored (NCT04474405 and NCT01992380) and non-Avid protocols and brought back to the clinic a minimum of 6 months after the initial flortaucipir PET scan for cognitive testing and an additional flortaucipir scan.
Groups:
- Cognitively Impaired: Clinically-diagnosed Alzheimer's disease (AD), mild cognitive impairment (MCI), and other dementing disorders (ODD) from the flortaucipir PET scan arm
- Healthy Volunteers: Male or female subjects ≥50 years of age without cognitive impairment from the flortaucipir PET scan arm
Period: Overall Study
Arm/Group | Cognitively Impaired | Healthy Volunteers
Started | 16 | 28
Completed | 16 | 21
Not Completed | 0 | 7
Not completed — Study terminated by sponsor | 0 | 7

BASELINE CHARACTERISTICS:
Population: Excluded 7 subjects who did not receive a flortaucipir scan
Groups:
- Cognitively Impaired: Clinically-diagnosed AD, MCI, and other dementing disorders (ODD) from the flortaucipir PET scan arm
- Healthy Volunteers: Healthy Volunteers from the flortaucipir PET scan arm
- Total: Total of all reporting groups
Arm/Group | Cognitively Impaired | Healthy Volunteers | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.15) | 75.3 (4.98) | 71.9 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 21 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 21 | 37
Amyloid status [Count of Participants; unit: Participants] — Amyloid status as previously determined either by PET imaging or cerebral spinal fluid (CSF) measures
  Participants
    Positive | 14 | 16 | 30
    Negative | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Tau Deposition
Description: Rate of tau deposition change as measured by flortaucipir standardized uptake value ratio (SUVr). For SUVr, a value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline scan and at least 6 months after baseline scan
Population: Amyloid positive and negative row n's reflect the subgroup counts.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | Cognitively Impaired | Healthy Volunteers
Number analyzed (Participants) | 16 | 21
standardized uptake value ratio (SUVr)
  Overall | 0.0347 (0.047) | -0.0008 (0.013)
  Amyloid Negative: number analyzed (Participants) | 2 | 5
  Amyloid Negative | 0.0364 (0.082) | -0.0026 (0.013)
  Amyloid Positive: number analyzed (Participants) | 14 | 16
  Amyloid Positive | 0.0345 (0.045) | -0.0002 (0.013)
Statistical Analysis 1: Comparison: Cognitively Impaired vs Healthy Volunteers; Overall change from baseline between groups. Test compared slopes of cognitively impaired (CI) vs healthy volunteers (HV). As the time between scans varied across subjects, an ANCOVA model was used to estimate slopes in each diagnosis group and test whether they were the different at 1 year. The flortaucipir change from baseline was used as the dependent variable in the model; Test type: Other; p = 0.2837, ANCOVA — Not adjusted for multiple comparisons. No a priori threshold was selected; Adjustments included baseline tau deposition, age, time (in years) between imaging, and included an interaction of time and enrolling diagnosis
Statistical Analysis 2: Comparison: Cognitively Impaired vs Healthy Volunteers; Change from baseline between groups for amyloid negative only. Test compared slopes of CI vs HV. As the time between scans varied across subjects, an ANCOVA model was used to estimate slopes in each diagnosis group and test whether they were different at 1 year. The flortaucipir change from baseline was used as the dependent variable in the model; Test type: Other; p = 0.9276, ANCOVA — Not adjusted for multiple comparisons. No a priori threshold was selected; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cognitively Impaired vs Healthy Volunteers; Change from baseline between groups for amyloid positive only. Test compared slopes of CI vs HV. As the time between scans varied across subjects, an ANCOVA model was used to estimate slopes in each diagnosis group and test whether they were different at 1 year. The flortaucipir change from baseline was used as the dependent variable in the model; Test type: Other; p = 0.6324, ANCOVA — Not adjusted for multiple comparisons. No a priori threshold was selected; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Administration of study drug until 48 hours post administration
Arm/Group | Cognitively Impaired | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/21
Other Adverse Events (participants affected / at risk) | 1/16 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitively Impaired (N=16) | Healthy Volunteers (N=21)
Headache (Nervous system disorders) | 1 (1) | NA — Moderate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data confidentiality for a period of 5 years following study termination